CLINICAL TRIAL: NCT01554046
Title: The Effect of Methylphenidate (Ritalin IR) Treatment in Familial Attention Deficit/Hyperactivity Disorder (ADHD)
Brief Title: The Effect of Methylphenidate Treatment in Familial Attention Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-12-8292-DG-CTIL
Record Dates: First submitted 2012-02-23; First posted 2012-03-14 (Estimated); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Attention Deficit/Hyperactivity Disorder Combined Type; ADHD Predominantly Inattentive Type; ADHD Predominantly Hyperactivity Type; ADHD-not Other Specified
Keywords: Attention Deficit Hyperactivity Disorder (ADHD); Methylphenidate- RITALIN IR (Immediate Release)
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- couples of first-degree family members (Experimental)
  Interventions: Drug: Methylphenidate- Ritalin IR (Immediate Release)

INTERVENTIONS:
Drug: Methylphenidate- Ritalin IR (Immediate Release) — Duration of treatment- 4 weeks. Dosage- up to 3 times/day.
  * Ages 6-12, up to 25Kg - 35mg maximum per day.
  * Ages 6-12, above 25Kg - 50mg maximum per day.
  * Ages 12-65, above 25Kg - 80mg maximum per day.

SUMMARY:
The purpose of this study is to investigate the familial response to Methylphenidate treatment (Ritalin IR) in two aspects: ADHD symptom's improvement and side-effects development.

DETAILED DESCRIPTION:
Attention Deficit/Hyperactivity Disorder (ADHD) is very prevalent and tends to continue from childhood to adult life. It's heritability is 76%. It was found that there is a greater ADHD prevalence in first-degree families of ADHD subjects- 4-6 times more than the general population.

Pharmacological treatment is the first line treatment today in ADHD, in children and adults, and Methylphenidate (specially Ritalin IR) is the first medication given for the disorder.

The study includes couples of first-degree family members, both diagnosed with ADHD. Subjects will receive Ritalin IR for 4 weeks and undergo several psychiatric and cognitive questionnaires at each time of the follow-up meeting (a total of 3).

ELIGIBILITY:
Inclusion Criteria:

* couples of first-degree family members, both diagnosed with ADHD (any type or ADHD-NOS) and need medical treatment.

Exclusion Criteria:

* subjects who receive other psychiatric medications: antipsychotic medications, antidepressants medications, anti-anxiety medications or mood stabilizers.
* people who suffer from psychotic disorder, bipolar disorder or other severe psychiatric disorders which are not stabilized.
* Alcohol/drugs addicted.
* people with chronic neurologic diseases.
* people with Autism or mental retardation.
* people with congenital heart defect.
* people with hypertension/tachycardia (>100 bpm).
* pregnancy or breast feed women.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-10; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression-Improvement scale | CGI scale score at 4 weeks <=2

SECONDARY OUTCOMES:
overall ADHD-Rating Scale (ADHD-RS) score | change from baseline in ADHD-RS at 2 weeks (reducing >30%), change from baseline in ADHD-RS at 4 weeks (reducing >30%)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Doron Gothelf, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- ADHD Medical Clinic, Child and Adolescent Psychiatry Unit, Sheba Medical Center, Ramat Gan, Israel